CLINICAL TRIAL: NCT05762159
Title: Analgesic Territory Assessment of the Spinal Erector Block Using Pupillometry
Acronym: TEASER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1272022/CHUSTE
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia, Local
Keywords: spinal erector block; pupillometry; loco-regional anesthesia; osteosynthesis
MeSH Terms: interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- erector spinae block: Patients receiving erector spinae block for pain management of spinal osteosynthesis. Pupillometer will be realized during analgesia (usual practice).
  Interventions: Other: data collected

INTERVENTIONS:
Other: data collected — data collected:
  * Morphological data of the patients
  * Data of the erector block realization
  * Pupillometric data :the variation of the pupil size on stimulation (in percentage of the base diameter)

SUMMARY:
Few works have studied the area of analgesia covered by the spinal erector block in an objective manner, especially on the cephalo-caudal spread. The available data are dissection works or subjective data such as thermoalgesic or epicritic sensitivity.

This information would however be relevant in order to propose a better analgesia. Indeed, it could explain certain failures by insufficient diffusion of the block. The use of a multistage block could be relevant, especially in the case of osteosynthesis on several vertebral levels.

DETAILED DESCRIPTION:
Pupillometry makes possible to monitor analgesia based on the pupillary dilation reflex to pain. The goal is to establish an objective mapping of these type of analgesia from these data.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving erector spinae block for pain management of spinal osteosynthesis

Exclusion Criteria:

* Patient refusal
* Known allergy to local anesthetics
* Contraindication to locoregional anesthesia (haemostasis disorder, infection, peripheral neuropathy)
* Technical impossibility to perform a spinal erector block
* Pathology with dysautonomia altering the pupillary reflex: diabetes mellitus with diabetic retinopathy, multiple sclerosis, systemic amyloidosis, uncontrolled hypertension, glaucoma
* Current treatment likely to alter pupillary dilation reflex to pain : antiemetic (droperidol, metoclopramide), alpha-2 agonist (clonidine)
* Serious psychiatric history
* Drug abuse
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving erector spinae block for pain management of spinal osteosynthesis will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
variation of the pupil size (in percentage) | During the surgery
  Evaluation the territory covered by the spinal erector block by variation of the pupil size (in percentage).
  Variation of the pupil size on stimulation will allow to deduce if the dermatome is covered by the spinal erector block analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Wodey, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No